CLINICAL TRIAL: NCT05964569
Title: Prospective Phase II Trial to Assess Feasibility of Individualized, Model-guided Optimization of Proton Beam Treatment Planning in Patients With Low Grade Glioma Multicentric, Prospective Interventional, Randomized, Observer Blind Two Arm (Active Control), Parallel Group Investigator-initiated Phase II Trial
Brief Title: Feasibility of Individualized, Model-guided Optimization of Proton Beam Treatment Planning in Patients With Low Grade Glioma
Acronym: INDIGO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Department Head, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RadOnk-Indigo
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Low Grade Glioma

STUDY DESIGN:
Intervention Model Description: randomized, observer blind two arm (active control), parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment plan (Active Comparator): Model-based NTCP is calculated after plan approval, however, no further adjustments are to be made to the approved treatment plan
  Interventions: Other: standard treatment plan, no optimization
- Optimized treatment plan (Experimental): Allocated to Control Calculation of normal tissue complication probability (NTCP) Model-guided replanning. Replanning is performed with Raysearch Raystation. Optimizations objectives are:
  1. the optimization objectives that control the maximum dose in the target volume employ a variable, LETd-dependent model for RBE that allows us to include the RBE-variations predicted by the NTCP model
  2. the periventricular volume, defined as the volume closer than 4 mm to the ventricular wall, is included into the optimization with a constraint on its Equivalent Uniform Dose (EUD) and with the variable RBE model described above. Thereby, the combined effect of the RBE variation and increased sensitivity of the periventricular volume, as predicted by the NTCP model, is included.
  The effectiveness of the re-planning is verified by a second NTCP computation.
  Interventions: Other: model-guided optimization of treatment plan

INTERVENTIONS:
Other: model-guided optimization of treatment plan — original treatmant plans are optimized based on model-based NTCP
  Arms: Optimized treatment plan
Other: standard treatment plan, no optimization — original treatment plans are not optimized
  Arms: Standard treatment plan

SUMMARY:
Low-grade glioma (LGG) represent typically slowly growing primary brain tumors with world health organization (WHO) grade I or II who affect young adults around their fourth decade. Radiological feature on MRI is a predominantly T2 hyperintense signal, LGG show typically no contrast uptake. Radiotherapy plays an important role in the treatment of LGG. However, not least because of the good prognosis with long term survivorship the timing of radiotherapy has been discussed controversially. In order to avoid long term sequelae such as neurocognitive impairment, malignant transformation or secondary neoplasms initiation was often postponed as long as possible

DETAILED DESCRIPTION:
Since patients with low grade glioma are expected to become long-term survivors, the prevention of long-term sequelae is particularly important. In addition to disease progression, also treatment related side effects such as decline of neurocognitive function, endocrine impairment or sensorineural deficits can have a negative impact on patient's quality of life.

Owing to the biophysical properties of protons with an inverse depth dose profile compared to photons and a steep dose fall of to the normal tissue, there is a strong rationale for the use of PRT in the treatment of patients with low-grade glioma. Although data from large randomized trials are still missing there is increasing evidence from smaller prospective trials and retrospective analyses that the expected advantages indeed transform into clinical advantages.

However, in about 20 % of all patients, late contrast-enhancing brain lesions (CEBL) appear on follow-up MR images 6 - 24 months after treatment. At HIT in Heidelberg and at OncoRay in Dresden, CEBLs have been observed to occur at very distinct locations in the brain and relative to the treatment field. Retrospective analysis has elucidated potential key factors that lead to CEBL occurrence. However, avoidance of CEBLs is hardly feasible using conventional treatment planning strategies. Model-aided risk avoidance denotes the use of model-based CEBL risk calculations as an auxiliary tool for clinical treatment planning: Model-based risk calculations and risk reduction via software-based optimization help the clinician to minimize risk of CEBL occurrence during treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* histologically proven low-grade glioma
* indication for definitive or adjuvant radiotherapy
* ability to understand character and personal consequences of the clinical trial
* written informed consent

Exclusion Criteria:

* previous cerebral irradiation
* contraindication for contrast-enhanced MRI
* neurofibromatosis
* participation in another clinical trial with competing objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2028-11-11 (Estimated)

PRIMARY OUTCOMES:
incidence of contrast enhancing brain leasions | observed within 24 months after PRT measured by quarterly contrast enhanced MRI of the brain
  the cumulative incidence of contrast enhancing brain lesions

SECONDARY OUTCOMES:
radiation-induced brain injuries | observed within 24 months after PRT measured by quarterly contrast enhanced MRI of the brain
  incidence of radiation-induced brain injuries > CTC°II
progression-free survival | observed within 24 months after PRT measured by quarterly contrast enhanced MRI of the brain
  number of surviving patients without tumor progression
overall survival | observed within 24 months after Proton Beam Therapy (PRT) measured by quarterly contrast enhanced MRI of the brain
  number of surviving patients
patient reported outcome | up to 24 months after completion of radiotherapy
  patient reported outcome according to points on the PRO-CTCAE questionaire, scored 0/1 for absent/present)
quality of life QLQ-C30 | up to 24 months after completion of PRT
  scores on the QLQ-C30 questionare, scored 0 (absence) to 5 (fully present)
quality of life QLQ-BN20 | up to 24 months after completion of PRT
  scores on the QLQ-BN20 questionare, scored 0 (absence) to 5 (fully present)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05964569/Prot_000.pdf